CLINICAL TRIAL: NCT04702308
Title: The Use of Non-Interruptive Alerts for Improving the Use of Clinical Decision Rules in the Emergency Department: A Cluster Randomized Controlled Trial
Brief Title: Non-Interruptive Alerts for Improving Use of Clinical Decision Rules
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Keaton Morgan, Postdoctoral Fellow, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 00137874
Record Dates: First submitted 2021-01-04; First posted 2021-01-08 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Pulmonary Embolism; Deep Vein Thrombosis; Minor Head Injury; Chest Pain; Neck Trauma
Keywords: clinical decision support; clinical decision rules
MeSH Terms: conditions — Pulmonary Embolism; Venous Thrombosis; Craniocerebral Trauma; Chest Pain

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention will contain two components: 1) a non-interruptive best practice advisory (BPA) in the Epic Storyboard and 2) a default suggested calculator tab in the MDCalc Connect app. Six clinical decision rules will be included: Canadian CT Head Rule, Canadian C-spine Rule, HEART Score, PERC Rule, Wells' PE Criteria and Wells' DVT Criteria. Predefined criteria based on chief complaint, patient age and vital signs will be used to determine when a decision rule may be relevant in a patient encounter. When a patient meets all of the predefined criteria, the intervention will be triggered.
  Interventions: Other: Clinical Decision Rule Alerts
- Control Group (No Intervention): The control group will be usual care. Specifically, providers in the control group will not receive the clinical decision rule alert or the default suggested calculator tab in the MDCalc Connect app. The control group providers will have access to the MDCalc Connect app in its standard form and functionality.

INTERVENTIONS:
Other: Clinical Decision Rule Alerts — The
  Arms: Intervention Group

SUMMARY:
This study is an extension of a planned quality improvement project that aims to promote standard of care by increasing the use of evidence-based clinical decision rules amongst emergency medicine providers in the University of Utah Emergency Department. Patient-specific information from the EHR will be used to recommend the use of relevant clinical decision rules to emergency medicine providers at the point-of-care. These recommendations will be in the form of non-interruptive alerts with one-click access to the suggested decision rules through the MDCalc Connect EHR add-on application. Specific aims of the study are to determine if 1) patient-specific non-interruptive alerts increase the use of clinical decision rules amongst emergency medicine providers and 2) an increase in the use of clinical decision rules affects provider ordering habits.

ELIGIBILITY:
Patient Inclusion Criteria:

* 16 years of age or older
* Qualifying chief complaint*

Patient Exclusion Criteria:

* None

  * A full list of the qualifying chief complaints is provided in Appendix A of the full research protocol.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2022-11-04 (Actual)

PRIMARY OUTCOMES:
Total clinical decision rule usage | During the intervention
  Composite measure of total number of clinical decision rules used through the MDCalc Connect app.

SECONDARY OUTCOMES:
Individual clinical decision rule usage | During the intervention
  Number of uses of individual clinical decision rules measured through the MDCalc Connect app.
Computed tomography pulmonary angiography studies | During the intervention
  The total number of computed tomography pulmonary angiography studies ordered
Computed tomography head studies | During the intervention
  The total number of computed tomography head without contrast studies ordered
Computed tomography c-spine studies | During the intervention
  The total number of computed tomography c-spine without contrast studies ordered
Lower extremity ultrasound | During the intervention
  The total number of lower extremity ultrasound studies ordered
d-dimer tests | During the intervention
  Total number of d-dimer blood tests ordered
Delta troponin tests | During the intervention
  Total number of times two or more troponin tests were ordered
Emergency department bounceback rate. | Up to 30 days after the intervention
  30-day emergency department return visit (or "bounceback") rate
Admission rate | During the intervention
  Hospital admission rate

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-17): https://cdn.clinicaltrials.gov/large-docs/08/NCT04702308/Prot_SAP_000.pdf